CLINICAL TRIAL: NCT02375282
Title: Physical and Functional Recovery From Cardiac Surgery in Hospitalized Patients: A Feasibility Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: Springfield College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BH-14-169
Record Dates: First submitted 2015-01-27; First posted 2015-03-02 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Coronary Artery Disease; Mitral Valve Insufficiency; Aortic Valve Stenosis; Aortic Valve Regurgitation; Mitral Valve Stenosis; Coronary Artery Bypass Graft Triple Vessel
Keywords: ambulation; cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Mitral Valve Insufficiency; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambulation Orderly Intervention (Experimental): Patients that are in this group are those randomized to receive visits from the ambulation orderly (ambulation group). The patients in this group will receive the visits from the ambulation orderly in addition to the standard of care that occurs with the rest of the hospital and with the control group.
  Interventions: Procedure: Ambulation orderly
- Control Group (No Intervention): This is for the patients who are randomized to receive the standard care of Baystate Medical Center. The standard of care will be nurse-directed ambulation, as is currently done in all other nursing floors at Baystate Medical Center. Nurses will be instructed to walk with the patients as they did before the initiation of the ambulation orderly and as they do when the orderly is on vacation, at conferences, training, or away for illness. These patients will not receive visits from the ambulation orderly.

INTERVENTIONS:
Procedure: Ambulation orderly — The responsibility of the ambulation orderly is to walk patients after having a cardiac surgery, such as a coronary artery bypass surgery or a valve surgery. Baystate Medical Center hired an ambulation orderly May 8, 2013. The ambulation orderly is generally a high school graduate with some training in safe lifting and exercise, but extensive training is not required. In general, the goal is to have 1 ambulation orderly present 7 days a week for 8 hr per day. When available, ambulation orderlies are responsible for walking the patients who have been cleared by the clinical exercise physiologist or nurse up to 4 times per day. The walking of the patients occurs through the halls of the 6th floor of the Mass Mutual wing of Baystate Medical Center.
  Arms: Ambulation Orderly Intervention

SUMMARY:
Ambulation following surgery has been found to be beneficial for patients; however, nurses and doctors struggle with getting post-operative, hospitalized patients to walk on their own. One promising strategy to address this might be an ambulation orderly, an employee whose single responsibility is to assure that patients walk 3-4 times per day. However, the effect of the ambulation orderly on post-operative physical activity has not yet been described. It is important to quantify what the ambulation orderly does in order to assess if this is an effective method for helping patients walk. As a result, the investigators will perform a pilot randomized controlled trial to test the effects of an ambulation orderly in patients hospitalized with recent cardiac surgery. Half of the patients will be assigned to walk with the ambulation orderly 3-4 times/day and the control group will be given standard nursing encouragement and assistance and encouragement to walk. The investigators will evaluate the average total daily step counts (over the hospital course, usually 4-7 days) and the change in walking distance between a baseline and a final 6 minute walk test. The investigators will also evaluate exercise physiologic parameters (heart rate, oxygen saturation) during ambulation, patient functional independence, and patient satisfaction.

DETAILED DESCRIPTION:
The investigators will perform a prospective randomized controlled trial at Baystate Medical Center, a 684-bed academic teaching hospital that serves as the referral center for a population of approximately 800,000 people living in Western Massachusetts.

The responsibility of the ambulation orderly is to walk patients after having a cardiac surgery, such as a coronary artery bypass surgery or a valve replacement or repair. Patients will be randomized to receive visits from the ambulation orderly (ambulation group) or to receive the standard care of Baystate Medical Center (control group). The standard of care will be nurse-directed ambulation, as is currently done in all other nursing floors at Baystate Medical Center. Nurses will be instructed to walk with the patients as they did before the initiation of the ambulation orderly and as they do when the orderly is on vacation, at conferences, training, or away for illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a cardiac surgery procedure (coronary artery bypass grafting surgery or valve surgery). Must be ambulatory prior to surgery

Exclusion Criteria:

* Unable to consent, cognitively impaired, and patients unable to walk prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Average Daily Step Counts while on M6 (cardiac surgery general floor.) | From arrival on M6 to hospital discharge. This is typically from post operative day 3 until post operative day 9-12.
  The patient will wear an accelerometer, which will keep track of the amount of steps the patient took each day over the course of the hospitalization.
Average change in walking distance between baseline and final 6-minute walk | From arrival on M6 (baseline) to hospital discharge (final). This is typically from post operative day 3 until post operative day 9-12
  Each patient will complete a 6 minute walk after arriving on M6 (from intensive care until) and again at hospital discharge. The difference in distance walked will be compared.

SECONDARY OUTCOMES:
Average Slope of Progression in Average Total Daily Step Counts | From arrival on M6 to hospital discharge. This is typically from post operative day 3 until post operative day 9-12.
  The patient will wear an accelerometer, which will keep track of the amount of steps the patient took each day. The progression between groups will be compared.
Average Daily Step Count on the 3rd day after arrival on M6 | 3rd day on M6 as part of study (typically post operative day 6 or 7)
  The step counts on the 3rd day after arrival on M6 will be compared in all groups. All patients are expected to still be in the hospital at this time.
Average Total Daily Energy Expenditure | From arrival on M6 to hospital discharge. This is typically from post operative day 3 until post operative day 9-12.
  The patient will wear an accelerometer, which will keep track of the total daily expenditure in calories per day.
Average Total Time in Activity | From arrival on M6 to hospital discharge. This is typically from post operative day 3 until post operative day 9-12.
  The patient will wear an accelerometer, which will keep track of the total time in activity.
Pre and post 6 minute walk test vital signs | Each time the 6 minute walk test is done.
  Heart rate, oxygen saturation, rating of perceived exertion, and rating of dyspnea will be measured before and after each 6 minute walk test.
Barthel Index | From arrival on M6 to hospital discharge. This is typically from post operative day 3 until post operative day 9-12.
  The research staff and nurses or exercise physiologist will complete a survey to assess the physical independence of the patients.
Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey | Following the hospital stay within 2-6 weeks
  The HCAHPS survey will be given to each patient at discharge to mail back to assess the overall satisfaction in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lindenauer, MD, MSc, Study Director — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Background] Brown CJ, Williams BR, Woodby LL, Davis LL, Allman RM. Barriers to mobility during hospitalization from the perspectives of older patients and their nurses and physicians. J Hosp Med. 2007 Sep;2(5):305-13. doi: 10.1002/jhm.209. PMID 17935241
- [Background] Callen BL, Mahoney JE, Grieves CB, Wells TJ, Enloe M. Frequency of hallway ambulation by hospitalized older adults on medical units of an academic hospital. Geriatr Nurs. 2004 Jul-Aug;25(4):212-7. doi: 10.1016/j.gerinurse.2004.06.016. PMID 15311196
- [Background] Pashikanti L, Von Ah D. Impact of early mobilization protocol on the medical-surgical inpatient population: an integrated review of literature. Clin Nurse Spec. 2012 Mar-Apr;26(2):87-94. doi: 10.1097/NUR.0b013e31824590e6. PMID 22336934
- [Derived] Pack QR, Woodbury EA, Headley S, Visintainer P, Engelman R, Miller A, Riley H, Lagu T, Lindenauer PK. Ambulation Orderlies and Recovery After Cardiac Surgery: A Pilot Randomized Controlled Trial. J Clin Exerc Physiol. 2017 Sep;6(3):42-49. doi: 10.31189/2165-6193-6.3.42. PMID 30687584